CLINICAL TRIAL: NCT02624570
Title: An Open-label, Multi-center, Expanded Treatment Protocol of Midostaurin (PKC412) in Adult Patients With Newly Diagnosed Fms-like Tyrosine Kinase Receptor (FLT3) Mutated Acute Myeloid Leukemia (AML) Who Are Eligible for Standard Induction and Consolidation Chemotherapy.
Brief Title: Midostaurin Access Program for Newly Diagnosed FLT3 (ITD or TKD) Mutated AML Adult Patients Eligible for Standard Induction and Consolidation Chemotherapy
Acronym: AMLFLT3
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CPKC412AUS56X
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia (AML) With; FLT3 Mutation, Internal Tandem Duplication (ITD) or Tyrosine Kinase Domain (TKD)
Keywords: AML; FLT3; ITD; TKD; acute myeloid leukemia; induction; consolidation; continuation; EAP; ETP; midostaurin; PKC412
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Midostaurin — Midostaurin, also known as PKC412 is a multi-kinase inhibitor of FLT3 (fms-like tyrosine kinase-3)
  Other Names: PKC412

SUMMARY:
The purpose of this study is to provide access to Midostaurin and gather additional safety data on the combination of Midostaurin and standard of care for adult patients with newly diagnosed Fms-like tyrosine kinase receptor (FLT3) mutated Acute Myeloid Leukemia (AML) who are eligible for standard induction and consolidation chemotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to provide Midostaurin (study drug) treatment to newly diagnosed FLT3 mutated (ITD or TKD) AML adult patients (18 years or older) eligible for standard standard induction (cytarabine + daunorubicin/Idarubicin) and consolidation (cytarabine) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained prior to any screening procedures. Patients must meet all Inclusion Criteria:

* Patient is able to communicate well with the investigator, to understand and comply with the requirements of the study.
* Patients must be 18 years of age or older; elderly patients must be fit to receive intensive induction and consolidation chemotherapy
* Patients must have a documented FLT3 mutation (ITD or TKD)
* Patients must have an ECOG Performance Status of ≤ 2
* Patients must have a documented unequivocal diagnosis of AML according to WHO 2008 classification (>20% blasts in the bone marrow and/or peripheral blood), excluding M3 (acute promyelocytic leukemia).
* Patients requiring intrathecal chemotherapy must have a minimum washout of 48 hours prior to the first dose of midostaurin
* AML patients with a history of antecedent treatment for myelodysplasia (MDS), e.g. azacitidine or decitabine, remain eligible for treatment on this study. These agents must have been discontinued for a period of at least 30 days or 5 half-lives of the drug (whichever is greater) before midostaurin can be administered.
* Secondary AML, e.g. patients with antecedent history of treatment for prior malignancy Patients must have the following laboratory values (Direct Bilirubin ≤ 2.5 x ULN, Serum Creatinine ≤ 2.5 x ULN)

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Prior therapy for AML with the following exceptions: (emergency leukapheresis, emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 5 days, cranial RT for CNS leukostasis (one dose only), growth factor/cytokine support)
* Patients with LVEF less than 45% (by echocardiogram or MUGA) or symptomatic congestive heart failure, Class III or IV according to New York Heart Association (NYHA) classification
* Patients with any uncontrolled illness, including, but not limited to, acute or chronic pancreatitis or uncontrolled infection
* QTc >500 msec on screening ECG. History of hypersensitivity to any drugs or metabolites of similar chemical classes as the IMP.
* Participation in a prior investigational interventional (drug) study with administration of the investigational product within 30 days or 5 half-lives of the investigational product, whichever is longer.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods.
* Sexually active males should not father a child during this study and for upto 5 months following.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - The Jordan Research and Education Center ABSMC Comprehensive Cancer Ctr, Berkeley, California
  - City of Hope National Medical Center Department of Hematology & HCT, Duarte, California
  - St. Judes Medical Center, Fullerton, California
  - University of Calif Irvine Medical Center Family Comp Cancer Cntr, Orange, California
  - Kaiser Permanente Northwest Kaiser, Denver, Colorado
  - Poudre Valley Hospital Poudre Valley Hospital -U of C, Fort Collins, Colorado
  - Memorial Healthcare System Memorial Healthcare System, Hollywood, Florida
  - UF Health Cancer Center at Orlando Health Orlando Health, Orlando, Florida
  - H Lee Moffitt Cancer Center and Research Institute SC - 5, Tampa, Florida
  - Augusta University Georgia Cancer Center Pharmacy, Augusta, Georgia
  - Rush University Medical Center Dept.of Rush UniversityMedCtr., Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana Blood and Marrow Institute Indiana Blood and Marrow Trans, Beech Grove, Indiana
  - Ft Wayne Medical Oncology and Hematology Inc, Fort Wayne, Indiana
  - Norton Cancer Institute Norton Cancer Institute, Louisville, Kentucky
  - University of Louisville / James Graham Brown Cancer Center Louisville 529-539, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute Harper Hosp. Invest. Pharmacy, Detroit, Michigan
  - Henry Ford Hospital SC, Detroit, Michigan
  - Mayo Clinic Mayo Clinic, Rochester, Minnesota
  - Nebraska Cancer Specialist/Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Healthcare Partners Medical Group, Las Vegas, Nevada
  - Weill Cornell Medical College NY Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center Univ of Rochester (7), Rochester, New York
  - Kaiser Permanente NW Region Kaiser Permanente Northwest, Clackamas, Oregon
  - Penn State University / Milton S. Hershey Medical Center Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center University of Pen/Abr Canc ctr, Philadelphia, Pennsylvania
  - Medical University of South Carolina Hematology-Oncology Division, Charleston, South Carolina
  - Erlanger Medical Center Erlanger Health System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Clinical Trials Center Division Hematology/Oncology, Nashville, Tennessee
  - University of Texas Medical Branch University of Texas MB, Galveston, Texas
  - McGovern Medical School at the University of Texas Health, Houston, Texas
  - Oncology Consultants Oncology Consultants, Houston, Texas
  - Methodist Healthcare System, San Antonio, Texas
  - Intermountain Healthcare - Huntsman Cancer Clinics Intermountain Healthcare (2), Murray, Utah
  - Huntsman Cancer Institute Univ of Utah, Salt Lake City, Utah
  - Virginia Oncology Associates Virginia Oncology Assoc. (6), Norfolk, Virginia
  - Swedish Cancer Institute Cancer Institute, Seattle, Washington
  - Veterans Affairs Puget Sound Health Care System VAMC Seattle, WA Divison, Seattle, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Cheyenne Regional Medical Center, Cheyenne, Wyoming

REFERENCES:
- [Derived] Roboz GJ, Strickland SA, Litzow MR, Dalovisio A, Perl AE, Bonifacio G, Haines K, Barbera A, Purkayastha D, Sweet K. Updated safety of midostaurin plus chemotherapy in newly diagnosed FLT3 mutation-positive acute myeloid leukemia: the RADIUS-X expanded access program. Leuk Lymphoma. 2020 Dec;61(13):3146-3153. doi: 10.1080/10428194.2020.1805109. Epub 2020 Aug 19. PMID 32812818